CLINICAL TRIAL: NCT01181986
Title: Exenatide and Postprandial Endothelial Dysfunction: Effects and Mechanisms
Brief Title: The Study of Exenatide Action on Vessel Function in Type 2 Diabetes and Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Collaborators: American Diabetes Association (Other); Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Juraj Koska, Research Health Scientist, Carl T. Hayden VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1-10-CT-31
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus, Impaired glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Exenatide; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide SC (Sub-study 1) (Experimental): Study groups will be individuals with recent onset (<3 years) or established (>5 years) T2D. The plan is to achieve 40 complete studies of subcutaneous injection of exenatide BID (Byetta®, 5 or 10 µg) or identically looking Placebo SC for 10 days, separated by 14-day washout period. On the next day after each treatment phase, a single dose of the assigned medication will be injected just before a fat-enriched breakfast meal. A lunch meal of similar caloric and nutrient content will be administered 4 hours following the breakfast meal. Endothelial function will be measured just prior to the injection and every 2 hours during 8-hour post-breakfast period.
  Interventions: Drug: Exenatide SC; Drug: Placebo SC
- Exenatide IV (Sub-study 2) (Experimental): Study group will be individuals with recent onset (<1 year) T2D on diet and impaired glucose tolerance. The plan is to achieve 35 complete studies. The intervention will include 3 randomly ordered visits with intravenous infusion of exenatide in the presence (v1) or absence (v2) of GLP-1 receptor inhibitor exendin-9, and a control test with Placebo IV without exendin-9 (v3). Endothelial function will be measured at baseline and 2 hours later during the final 15 minutes of the infusion cocktails. Study participants will remain fasting during the test visit (3 hours total).
  Interventions: Drug: Exenatide IV; Drug: Exendin-9; Drug: Placebo IV

INTERVENTIONS:
Drug: Exenatide SC — Exenatide 5-10 ug sc BID/10 days
  Other Names: Byetta, exendin-4
  Arms: Exenatide SC (Sub-study 1)
Drug: Exenatide IV — 50 ng/min intravenously for 45 minutes on 2 out of 3 study visits separated by 5-10 days
  Other Names: exendin-4, Byetta
  Arms: Exenatide IV (Sub-study 2)
Drug: Placebo SC — Placebo sc BID/10days
  Other Names: placebo
  Arms: Exenatide SC (Sub-study 1)
Drug: Exendin-9 — Primed (6,000 pM/kg), continuous (600 pM/kg) intravenous infusion for 75 minutes on 1 out of 3 study visits.
  Other Names: exendin-(9-39)
  Arms: Exenatide IV (Sub-study 2)
Drug: Placebo IV — Intravenous infusion for 45 minutes on 1 out of 3 visits
  Other Names: placebo
  Arms: Exenatide IV (Sub-study 2)

SUMMARY:
The purpose of this investigation is to evaluate whether exenatide, a type 2 diabetes medication, will improve the function of the innermost part of the arterial wall called the endothelium after a fat-enriched meal and to determine how this occurs. The results of this study will help to determine and understand a novel action of this group of diabetes medications based on the action of naturally occuring gut substances called incretins. This may have a significant impact on cardiovascular health in patients with early and longstanding diabetes.

DETAILED DESCRIPTION:
Two independent, double-blinded, crossover substudies will be conducted to test the effect of exenatide on daylong post-meal and fasting endothelial function. We will measure endothelial function measured by peripheral arterial tonometry (EndoPAT2000, Itamar Inc.). Patients with recent onset (<3 years) or established (>5 years, Substudy 1 only) diabetes and impaired sugar tolerance (Substudy 2 only) will be studied. The plan is to complete studies in 75 patients (40 in Substudy 1 and 35 in Substudy 2).

In Substudy 1 patients will get twice a day a skin injection of exenatide (Byetta) or identically looking placebo for 10 days, separated by 14-day period. On the next day after each treatemnt period (day 11), they get just one injection and eat a fat-enriched breakfast. A fatty lunch of similar caloric content will be given 4 hours following the breakfast. Endothelial function will be measured just prior to the injection and every 2 hours for total 8 hours.

In Substudy 2, patients on 3 different days will get infusion of exenatide withg or without a blocking drug exendin-9, and a control test with placebo without exendin-9. Endothelial function will be measured before the infusion and 2 hours later during the final 15 minutes of the infusion cocktails. Patients will not eat any meal during the test visits.

ELIGIBILITY:
Inclusion Criteria:

* US Veterans
* type 2 diabetes mellitus (T2D) diagnosed within 3 years with good glycemic control on diet, metformin, or sulfonylurea agents or combinations of these agents (HbA1c ≤8.0%)
* T2D diagnosed ≥ 5 years prior to study enrollment
* Impaired glucose tolerance

Exclusion Criteria:

* T2D not meeting inclusion above criteria for duration of diabetes or HbA1c values
* known or suspected T1D (early onset age, low body mass index, lack of family history)
* TZD use in the prior 3 months
* prior regular use of insulin
* Creatinine >2.0 mg/dl or other laboratory or clinical evidence of kidney disease
* anemia
* known active liver disease or hepatic enzyme elevation two-and-a half times above normal
* acute bacterial or viral illness or evidence of other active infection in the past 4 weeks
* stable or unstable angina or other major illness in the past 6 months
* Raynaud's disease or any rheumatic disease affecting fingers
* current regular use of anti-inflammatory medications or antioxidants, including over the counter medications and high dose salicylates (>1 g/day);
* subjects receiving lipid lowering or anti-hypertension medications must be on stable doses for at least 2 months prior to participation.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juraj Koska, MD, PhD, Principal Investigator — Phoenix VA Healthcare System
Locations (1):
- Phoenix VA Medical Center, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Then Placebo (Sub-study 1): Patients received exenatide 5-10 ug sc BID for 10 days. On day 11, after receiving AM dose, vascular and blood parameters responses to study meal were tested.
- Placebo Then Exenatide (Sub-study 1): Patients received placebo sc BID for 10 days. On day 11, after receiving AM dose, vascular and blood parameters responses to study meal were tested.
- Exenatide IV (Sub-study 2): Patients received in random order on single day an intravenous infusion of (1) Saline+Exenatide, (2) Exendin-9+Exenatide or (3) Saline+Placebo
Period: Phase 1
Arm/Group | Exenatide Then Placebo (Sub-study 1) | Placebo Then Exenatide (Sub-study 1) | Exenatide IV (Sub-study 2)
Started | 19 | 23 | 34
Saline+Exenatide | 0 (N/A for this arm) | 0 (N/A for this arm) | 32
Saline+Placebo | 0 (N/A for this arm) | 0 (N/A for this arm) | 33
Exendin-9+Exenatide | 0 (N/A for this arm) | 0 (N/A for this arm) | 33
Completed | 18 | 22 | 32
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Period: Phase 2
Arm/Group | Exenatide Then Placebo (Sub-study 1) | Placebo Then Exenatide (Sub-study 1) | Exenatide IV (Sub-study 2)
Started | 18 | 22 | 0 (N/A for Sub-study 2)
Completed | 18 | 18 | 0
Not Completed | 0 | 4 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Medical condition | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sub-study 1: Exenatide SC: Exenatide 5-10 ug or placebo sc BID/10 days, day 11 AM dose and meal test - crossover study
- Sub-study 2: Exenatide IV: Intravenous infusion of (1) Saline+Exenatide, (2) Saline+Placebo or (3) Exendin-9+Exenatide on 3 seperate days, crossover study
- Total: Total of all reporting groups
Arm/Group | Sub-study 1: Exenatide SC | Sub-study 2: Exenatide IV | Total
Number analyzed (Participants) | 42 | 34 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (6) | 60 (6) | 61 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 42 | 32 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 36 | 29 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33 (6) | 33 (12) | 33 (9)
Glycated hemoglobin [Mean (Standard Deviation); unit: %] | 6.6 (0.9) | 6.1 (0.5) | 6.4 (0.8)
Diabetes duration (years) [Median (Inter-Quartile Range); unit: years] | 6 [1 to 9] | 0 [0 to 1] | 6 [1 to 9]
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 128 (8) | 125 (12) | 127 (14)
Diastolic BP (mmHg) [Mean (Standard Deviation); unit: mmHg] | 78 (8) | 80 (8) | 79 (8)
History of hypertension [Number; unit: participants]
  Yes | 33 | 16 | 49
  No | 9 | 18 | 27
Lipid-lowering therapy [Number; unit: participants]
  Yes | 5 | 15 | 20
  No | 37 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Reactive Hyperemia Index (RHI)
Description: Greater RHI reflects greater endothelial function. It is calculated as average post-ischemia pulse magnitude divided by average pre-ischemia pulse magnitude. Results are expressed as least-square means of ANCOVA models.
Time Frame: 0, 2, 4, 6 and 8 hours on Day 11 (Sub-study 1); 0 and 120 minutes on test Days 1, 2 & 3 (Sub-study 2)
Measure: Least Squares Mean (Standard Error); unit: ratio
Groups:
- Exenatide (Subs-study 1): Exenatide: Exenatide 5-10 ug sc BID/10 days
- Placebo (Sub-study 1): Placebo sc BID for 10 days
- Saline+Exenatide (Sub-study 2): Infusion of saline (min 0-75), added exenatide infusion (min 30-75)
- Saline+Placebo (Sub-study 2): Infusion of saline (min 0-75), added placebo infusion (min 30-75)
- Exendin-9+Exenatide (Sub-study 2): Infusion of exendin-9 (min 0-75), added exenatide infusion (min 30-75)
Arm/Group | Exenatide (Subs-study 1) | Placebo (Sub-study 1) | Saline+Exenatide (Sub-study 2) | Saline+Placebo (Sub-study 2) | Exendin-9+Exenatide (Sub-study 2)
Number analyzed (Participants) | 36 | 36 | 32 | 32 | 32
ratio | 1.90 (0.005) | 1.79 (0.05) | 2.24 (0.07) | 1.95 (0.07) | 1.99 (0.07)
Statistical Analysis 1: Comparison: Exenatide (Subs-study 1) vs Placebo (Sub-study 1); Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for treatment sequence, group (diabetes duration) and time
Statistical Analysis 2: Comparison: Saline+Exenatide (Sub-study 2) vs Saline+Placebo (Sub-study 2); Test type: Superiority or Other; p = 0.006, ANCOVA; Adjusted for treatment sequence
Statistical Analysis 3: Comparison: Saline+Exenatide (Sub-study 2) vs Exendin-9+Exenatide (Sub-study 2); Test type: Superiority or Other; p = 0.003, ANCOVA; Adjusted for treatment sequence

2. Secondary Outcome: Plasma Triglycerides
Description: Triglycerides concentrations were measured before and 2, 4, 6 and 8 hours following study drug. Results are expressed as least-square means of ANCOVA models adjusted for sampling time and intervention sequence.
Time Frame: 0, 2, 4, 6 and 8 hours post-study drug on day 11
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Groups:
- Exenatide (Sub-study 1): Patients received exenatide 5-10 ug sc BID for 10 days. On day 11, after receiving AM dose, vascular and blood parameters responses to study meal were tested.
- Placebo (Sub-study 1): Patients received placebo sc BID for 10 days. On day 11, after receiving AM dose, vascular and blood parameters responses to study meal were tested.
Arm/Group | Exenatide (Sub-study 1) | Placebo (Sub-study 1)
Number analyzed (Participants) | 36 | 36
mg/dl | 175 (14) | 230 (14)
Statistical Analysis 1: Comparison: Exenatide (Sub-study 1) vs Placebo (Sub-study 1); Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for treatment sequence and diabetes duration group

3. Secondary Outcome: Plasma Glucose
Description: Plasma glucose was measured before and 2, 4, 6 and 8 hours following study drug administration. Results are expressed as least-square means of ANCOVA models adjusted for sampling time and intervention sequence.
Time Frame: 0, 2, 4, 6, and 8 hours post-study drug on day 11
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Exenatide (Sub-study 1) | Placebo (Sub-study 1)
Number analyzed (Participants) | 36 | 36
mg/dl | 115 (5) | 136 (5)
Statistical Analysis 1: Comparison: Exenatide (Sub-study 1) vs Placebo (Sub-study 1); Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Groups:
- Exenatide SC (Sub-study 1): Exenatide 5-10 ug sc BID/10 days, AM dose and meal test on day 11
- Placebo SC (Sub-study 1): Placebo sc BID/10days, AM dose and meal test on day 11
- Saline+Exenatide IV (Sub-study 2): Intravenous infusion of saline (min 0-75), added intravenous infusion of exenatide (min30-75)
- Saline+Placebo (Sub-study 2): Intravenous infusion of saline (min 0-75), added intravenous infusion of placebo (min30-75)
- Exendin-9+Exenatide IV (Sub-study 2): Intravenous infusion of exendin-9 (min 0-75), added intravenous infusion of placebo (min30-75)
Arm/Group | Exenatide SC (Sub-study 1) | Placebo SC (Sub-study 1) | Saline+Exenatide IV (Sub-study 2) | Saline+Placebo (Sub-study 2) | Exendin-9+Exenatide IV (Sub-study 2)
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/32 | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 16/41 | 3/41 | 0/32 | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Exenatide SC (Sub-study 1) (N=41) | Placebo SC (Sub-study 1) (N=41) | Saline+Exenatide IV (Sub-study 2) (N=32) | Saline+Placebo (Sub-study 2) (N=33) | Exendin-9+Exenatide IV (Sub-study 2) (N=33)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0/34 (0) | 0 (0) | 1 (1) | 0 (0) — The event occured 13 days after the test visit during which patient received intravenous infusion of saline with placebo. The event was considered unrelated to the study per IRB decision.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide SC (Sub-study 1) (N=41) | Placebo SC (Sub-study 1) (N=41) | Saline+Exenatide IV (Sub-study 2) (N=32) | Saline+Placebo (Sub-study 2) (N=33) | Exendin-9+Exenatide IV (Sub-study 2) (N=33)
Nausea (Gastrointestinal disorders) | 14 (14) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No